CLINICAL TRIAL: NCT01632410
Title: The Cardiac Autonomic Nervous System State and Response to Reflective, Motor and Cognitive Stimuli Among Patients Post Stroke: A Follow-up Study
Brief Title: The Autonomic Nervous System State and Response to Different Stimuli Among Patients Post Stroke: A Follow-up Study
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Sponsor
Other Study IDs: TASMAC-12-NB-0227-12-CTIL
Record Dates: First submitted 2012-06-20; First posted 2012-07-03 (Estimated); Last update posted 2012-07-03 (Estimated); Status verified 2012-06

CONDITIONS: Stroke
Keywords: autonomic nerve system; post stroke; focus of study: to describe the autonomic nerve system function post stroke; autonomic nervous system
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (5):
- Study group 1: Post hemispheral ischemic stroke cognitively intact. Exclusion: Subjects with severe visual or hearing impairments, stroke location brain steam.
  The group will be divided in to 4 goups acording to stroke specific location as demonstrated in MRI.
- Control: Control: Healthy subjects resemble in age and sex
- Study -3: As explained the subjects will be divided into 4 groups acording to the stroke location. this is in order to evaluat the relationship between location and autonomic responed.
- Stydy -2: As explained the subjects will be divided into 4 groups acording to the stroke location. this is in order to evaluat the relationship between location and autonomic responed.
- Stydy- 4: As explained the subjects will be divided into 4 groups acording to the stroke location. this is in order to evaluat the relationship between location and autonomic responed.

SUMMARY:
The study describes the autonomic control system function in subjects post stroke in comparison with healthy subjects.

Aims: To describe the Autonomic hart rate control system function in post stroke subjects in different rehabilitation levels in comparison with healthy subjects.

To examine the reflective reaction of the autonomic control system as reflected in the heart rate variability to stimulations subjects in different rehabilitation levels in comparison with healthy subjects.

To examine the autonomic control system reaction as reflected in the heart rate variability to physical and cognitive action subjects in different rehabilitation levels in comparison with healthy subjects.

DETAILED DESCRIPTION:
Subjects will be examined 3 times: a week 1 and 3 month post stroke. Control consist similar in description healthy subjects, will be examined once. Each test includes 24 hours Holter surveillance and an examine that include general check that reflects the autonomic reaction to different manipulation.

The examination description:

A. Prior to the examination subjects will be asked to fill the mRS, NIHSS forms.

B. Subjects will receive an examination that includes

* General neurological examination (strength, deep and superficial sensation, cognitive test and pain level.) C. Holter will be place for 24 hours. And autonomic examination test will be conducted
* Grip Test: emphases the sympathetic system.
* Breathing Test: emphases the parasympathetic system. D. Manipulation to examine the two sub systems. Each manipulation lasts1 minute.

ELIGIBILITY:
Inclusion Criteria:

* Post hemispheral ischemic stroke cognitively intact.

Exclusion Criteria:

* Subjects with severe visual or hearing impairments, stroke location brain steam.

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Post hemispheral ischemic stroke cognitively intact.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2012-07; Primary Completion 2012-11 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
RMSSD change | 3 month post stroke
  The root mean square successive difference (RMSSD) in heart period series is a time domain measure of heart period variability.
  we will follow up the change in RMSSD at 1st and 3rd month post stroke

SECONDARY OUTCOMES:
6mwt | 3 month post stroke
  Endurance will be measured with the 6 minute walk test (6MWT). we will follow up the endurane change.
Patient's characteristics | 3 month post stroke
  a. Patient's characteristics questionnaire will include data such as: age, gender, health condition, medication, habits, education, etc.
  B. mRS and NIHSS questionears

CONTACTS AND LOCATIONS:
Overall Officials: Nathan Borshtin, Prof., Principal Investigator — Tel Aviv Suraski medical center
Locations (1):
- Tel Aviv Souraski Medical Center Neurology department, Tel Aviv, Israel